CLINICAL TRIAL: NCT04342364
Title: Oocyte Survival After Vitrification With Slush Nitrogen Compared With Liquid Nitrogen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Reproductive Medicine Associates of New Jersey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: RMA-2020-02
Record Dates: First submitted 2020-04-08; First posted 2020-04-13 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2022-01

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial in a paired design
Who Masked: Outcomes Assessor
Masking Description: embryologist assessing oocyte survival (primary outcome) is blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Slush nitrogen (Active Comparator): oocytes are randomized to undergo vitrification utilizing slush nitrogen
  Interventions: Other: Vitrification via slush nitrogen
- Liquid Nitrogen (Active Comparator): oocytes are randomized to undergo vitrification utilizing liquid nitrogen which is the current standard of care
  Interventions: Other: Vitrification via liquid nitrogen

INTERVENTIONS:
Other: Vitrification via slush nitrogen — oocytes will be vitrified using slush nitrogen
  Arms: Slush nitrogen
Other: Vitrification via liquid nitrogen — oocytes will be vitrified using liquid nitrogen which is currently routine practice
  Arms: Liquid Nitrogen

SUMMARY:
The purpose of this study is to determine if the use of slush nitrogen results in higher post-thaw survival rates for oocytes compared to conventionally used liquid nitrogen.

DETAILED DESCRIPTION:
The study is a randomized, controlled trial which seeks to characterize oocyte survival rate following vitrification and subsequent warming with both slush nitrogen and liquid nitrogen. After warming, fertilization and embryology outcomes will be assessed.

Oocyte donors and a single donor sperm source will be utilized. Following enrollment, oocyte donors will undergo ovarian stimulation and oocyte retrieval. The mature (MII) oocytes obtained for each patient will then be assigned a number and randomized via block randomization to one of two treatment groups (liquid nitogen or slush nitrogen). Through block randomization, this will create a paired population of oocytes so that half of each patient's oocytes will undergo cryopreservation with liquid nitrogen and half will undergo cryopreservation with slush nitrogen. Timing of hyaluronidase stripping and vitrification will be consistent with current institutional clinical practice for oocytes.

Following cryopreservation, oocytes will be warmed and intracytoplasmic sperm injection will be performed and subsequent embryology outcomes tracked.

ELIGIBILITY:
Major Inclusion Criteria for oocyte donors:

1. Age 30 years or younger who meet institutional criteria to be an oocyte donor.
2. Patients who agree to donate oocytes for research purposes and agree to the study protocol.
3. The subgroup of oocyte donors age 35-38 will not be part of the primary analysis, and therefore will not be required to meet the age criteria listed above. The older group of donors will be chosen as the clinical discretion of the study investigators. No specific ovarian reserve cutoffs will be required, although factors related to ovarian reserve will be taken into consideration.

Major Exclusion Criteria for oocyte donors:

1. Under 18 years old
2. All patients who do not voluntarily give their written consent for participation.
3. Patients who do not meet standard institutional criteria for oocyte donation.
4. A diagnosis of polycystic ovarian syndrome (PCOS).

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2020-04-08 (Actual); Primary Completion 2021-05-11 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
oocyte survival rate | within 5 minutes post warming
  number of viable oocytes post warming

SECONDARY OUTCOMES:
fertilization rate | 18 hours post injection
  number of zygotes post intracytoplasmic sperm injection procedure
blastulation rate | 4-6 days after fertilization
  number of zygotes reaching the blastocyst stage of embryo development
euploid rate | 1 week after trophectoderm biopsy
  number of chromosomally normal embryos

CONTACTS AND LOCATIONS:
Locations (1):
- Reproductive Medicine Associates of New Jersey, Basking Ridge, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hanson BM, Kim JG, Suarez SI, Ackerman BK, Comito CE, Pangasnan R, Seli E, Hong KH, Scott RT Jr. Embryology outcomes after oocyte vitrification with super-cooled slush nitrogen are similar to outcomes with conventional liquid nitrogen: a randomized controlled trial. Fertil Steril. 2022 Jan;117(1):106-114. doi: 10.1016/j.fertnstert.2021.08.043. Epub 2021 Oct 13. PMID 34654569